CLINICAL TRIAL: NCT01690156
Title: Double Blinded Randomized Control Trial on the Effects of Ultrasound Probe Position on Ultrasound-guided Nerve Blocks
Brief Title: Trial on the Effects of Ultrasound Probe Position on Ultrasound-guided Nerve Blocks
Status: Terminated | Type: Observational
Why Stopped: This is not a clinical trial and was inadvertently entered in the system.
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Other Study IDs: Probeposition
Record Dates: First submitted 2012-09-17; First posted 2012-09-21 (Estimated); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: In-plane Ultrasound-guided Regional Anesthesia Performance
Keywords: In-plane; Ultrasound-guided regional anesthesia performance; Probe position; Needle visualization

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Parallel Probe Position: Performing the simulated interscalene block with the ultrasound probe parallel to the shoulders of the person performing the block
- Perpendicular Probe Position: Performing the simulated interscalene block with the ultrasound probe perpendicular to the shoulders of the person performing the block

SUMMARY:
Ultrasound has been used to guide a needle to inject local anesthetics around nerves. This is usually done in the same plane as the ultrasound beam in America and is known as an in-plane technique. When done correctly, the entire needle is visualized on the ultrasound screen as it approaches the nerves which are also seen on the same screen the entire time. The ultrasound probe can be held perpendicular or parallel to the shoulders of the person performing the in-plane technique. Our hypothesis is that holding the ultrasound probe perpendicular to the shoulder is superior to holding the probe parallel to the shoulder during an in-plane ultrasound guided regional anesthesia technique.

DETAILED DESCRIPTION:
Right handed volunteers with no prior exposure to ultrasound techniques are used in this study. They will be randomly assigned to be shown an instructional video on how to perform an in-plane ultrasound guided needling technique on a realistic simulation target. The two videos are identical with the exception of the probe position. A blinded assessor will time the volunteers performance behind a screen and note the duration in which the needle is not visualized in the ultrasound screen.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Right handed
* Aged 18 to 55

Exclusion Criteria:

* Any person who has prior knowledge about ultrasound imaging or regional anesthesia
* Any person who has prior experience with laparoscopy or biopsy
* Any person who has problems with depth of field or simple hand eye co-ordination task

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers naiive to ultrasound techniques
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Time taken to perform a simulated interscalene block | 1 hour
  Time taken to perform a simulated interscalene block after watching an instructional video on ultrasound guided regional anesthesia on the simulated targets

SECONDARY OUTCOMES:
Duration where the entire needle is not visualized when performing the simulated interscalene block | 1 hour
  Time taken to perform a simulated interscalene block after watching an instructional video on ultrasound guided regional anesthesia on the simulated targets

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas C Lam, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States